CLINICAL TRIAL: NCT05055583
Title: Toripalimab in Combination With Platinum-based Chemotherapy in Patients With Mutation-negative Stage IV Oligometastatic NSCLC: A Phase II Study.
Brief Title: Toripalimab in Combination With Platinum-based Chemotherapy for Mutation-negative Stage IV Oligometastatic NSCLC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tang-Du Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JS001-ISS-CO338
Record Dates: First submitted 2021-08-29; First posted 2021-09-24 (Actual); Last update posted 2021-09-24 (Actual); Status verified 2021-09

CONDITIONS: NSCLC Stage IV; Oligometastasis
Keywords: anti-PD-1; Toripalimab
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — toripalimab; Platinum Compounds

STUDY DESIGN:
Intervention Model Description: Single-arm, sigle-center, prospective phase II study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Toripalimab in Combination With Platinum-based Chemotherapy (Experimental): Participants receive totally 3-4 cycles of toripalimab combined with platinum-based chemotherapy neoadjuvant treatment during preoperative period. After the last treatment (Day 21 of Cycle 4), surgery will be performed within 4-6 weeks. Postoperatively, a comprehensive evaluation will be conducted by the investigator, and the intention was to receive maintenance therapy within 6-12 weeks of the MDT assessment.
  Interventions: Drug: Toripalimab in Combination With Platinum-based Chemotherapy; Procedure: Surgical treatment stage; Drug: Adjuvant treatment stage

INTERVENTIONS:
Drug: Toripalimab in Combination With Platinum-based Chemotherapy — Toripalimab will be administered at a fixed dose of 80 mg (2ml)/vial, IV, D1, with a full dose of 240 mg at one time, every 3 weeks for 3-4 cycles. Squamous cell carcinoma will be combined with cisplatin/carboplatin and Nab-paclitaxel: carboplatin, AUC=5, D1, IV, q3w, or cisplatin, 75 mg/m2, IV, q3w, and Nab-paclitaxel, 130 mg/m2, D1, IV, q3w, for 3-4 cycles. Non-squamous cell carcinoma will be combined with cisplatin/carboplatin and Pemetrexed, cisplatin/carboplatin is the same as above, Pemetrexed will be given at 500 mg/m2, D1, IV, q3w, for 3-4 cycles.
  Other Names: Toripalimab Injection; JS001; Teruipuli Dankang; TuoYI
Procedure: Surgical treatment stage — After the last treatment (Day 21 of Cycle 4), surgery was performed within 4-6 weeks.
Drug: Adjuvant treatment stage — Postoperatively, a comprehensive evaluation will be conducted by the investigator, and the intention will receive maintenance therapy within 6-12 weeks of the MDT assessment. Toripalimab: a fixed dose of 80 mg (2ml)/vial, IV, D1, a full dose of 240 mg at one time, every 3 weeks administered until PD or intolerable toxicity, for a maximum duration of 1 year.
  Other Names: Toripalimab Injection; JS001; Teruipuli Dankang; TuoYI

SUMMARY:
In recent years, immune checkpoint inhibitors targeting cytotoxic T-lymphocyte antigen-4, programmed death-1, and programmed death-ligand 1 have achieved milestones in the treatment of NSCLC, from back-line to first-line, and beyond. Is changing the standard of care for NSCLC. Currently, several phases Ⅲ clinical studies of neoadjuvant immunity combined with standard chemotherapy are underway, suggested that neoadjuvant ICI therapy is a promising way for locally advanced lung cancer. As an intermediate state in the process of tumor metastasis, Oligometastatic NSCLC patients have a better prognosis and more likely to benefit from local treatment than patients with extensive distant metastasis. However, there have been few reports of salvage surgery after ICI treatment in Oligometastatic NSCLC, and only one case has been reported to date. There is therefore a need to further gather evidence on salvage surgery after ICI.

DETAILED DESCRIPTION:
This is a single-center, single-arm, prospective phase II study to evaluate the efficacy and safety of toripalimab in combination with platinum-based and surgery in patients with mutation-negative stage IV Oligometastatic NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 ~ 70 years old, male or female.
* ECOG PS: 0 ~ 1. Patients with an ECOG score of 2 ~ 3 due to bone pain alone, assessed by the investigator, were allowed to be included.
* Histologically or cytologically confirmed stage IV Oligometastatic NSCLC (T1-3, N0-2, M1) according to The AJCC 8th edition TNM classification for lung cancer; The limitation of Oligometastatic was that the number of metastatic tumor foci ≤3 and only 1 organ was involved (excluding the primary organ). The involved metastatic organs were brain, liver, unilateral adrenal gland and bone.
* Proved EGFR, ALK, ROS1 wild-type non-small cell lung cancer.
* All patients should be evaluated by complete staging at baseline, and the confirmation of Qligometastases should include whole-body imaging (chest, abdominal, bone scan, or PET-CT).
* Patients with brain metastases who are assessed by adjuvant staging with PET-CT or magnetic resonance imaging (MRI) at baseline and who are expected to receive or have received radical treatment for the metastases (LAT), which is assessed and administered by the MDT team and includes surgery, radiation therapy, or a combination of both, Patients who have received treatment for intracranial lesions should have achieved neurological stability (other than residual signs or symptoms associated with CNS treatment) for at least 2 weeks, and at least 4 weeks after initial treatment with the treatment protocol in this study.
* Exist in patients with bone metastases, baseline imaging should be carried out in accordance with the requirements of this study confirmed that always happens skeletal related events (pathologic fracture, bone radiation, surgery, or spinal cord compression), 4 words patients in stable condition, before the start of the study were allowed in, but it must be submitted to the team before treatment and the current state of disease management, to ensure that qualified cases, Patients with bone metastases are allowed to receive bisphosphonates unless contraindicated or not recommended by the investigator.
* For patients with adrenal metastases, unilateral (non-primary) adrenal metastases should be confirmed by MRI or PET-CT at baseline and are expected to receive radical LAT therapy.
* For patients with liver metastases, patients at baseline should meet adequate or good liver function without hepatic encephalopathy or ascites, and are expected to receive radical/partial radical therapy for liver Oligomastatic lesions.
* Measurable target lesions were present at baseline according to RECIST 1.1 evaluation criteria.
* Vital organ function meets the following requirements (no blood components or cell growth factors are allowed to be used for 2 weeks prior to the start of study treatment)：

  1. blood routine:

     a) ANC ≥1.5×109/L; b) HB ≥9 g/dL; c) PLT ≥90×109/L; d) ALB ≥2.8 g/dL.
  2. Blood biochemistry:

     1. TBIL ≤1.5 ULN; b) ALT、AST≤2.5 ULN (If abnormal liver function is caused by oligosaccharide metastasis, ≤5.0 ULN); c) sCr≤1.5 ULN, Endogenous creatinine clearance rate ≥50ml/min (Cockcroft-Gault formula); d) BUN ≤ 2.5 ULN; e) Normal thyroid function (if TSH is not within the normal range at baseline, and if T3 and free T4 are within the normal range, then subjects will still meet the inclusion criteria).
* Expected survival ≥3 months.
* Fertile female subjects should conduct a urine or serum pregnancy test within 7 days prior to receiving the first study drug administration and prove negative and be willing to use an effective method of contraception during the study period until 12 months after the last study drug administration. For male subjects whose partners are women of reproductive age, effective contraception should be used during the trial and for 12 months after the last dosing.
* Patients voluntarily enrolled in this study and signed informed consent (ICF), with good compliance and follow-up.

Exclusion Criteria:

Subjects who meet any of the following criteria will be excluded from the study:

* Non-small cell lung cancer patients who do not meet the inclusion criteria for pathological types and primary sites of the lung.
* There are metastatic organs >1 kinds and metastatic lesions >3.
* Exact evidence confirms the presence of EGFR, ALK, ROS 1 gene mutations in non-small cell lung cancer.
* Have received systemic antitumor therapy or any other form of immune checkpoint inhibitor after diagnosis of stage IV Oligometastatic NSCLC.
* By MDT assessment, the primary lung lesion is expected to be inoperable, the primary tumor or metastases result in direct invasion or clinically highly suspected direct invasion of the main vascular wall, or the presence of malignant pleural or pericardial effusion.
* The Oligometastases were identified by the investigators as secondary primary tumors.
* Patients with brain metastases have proven to have CNS metastases and/or cancerous meningitis that, in the investigator's judgment, cannot be treated with radical treatment.
* Patients with bone metastases have demonstrated prior or current signs of osteoporosis/osteomyelitis of the jaw, or a history of uncontrolled osteoporosis fractures.
* Patients with liver metastases had hepatic encephalopathy in the past 6 months or clinically significant ascites at study enrollment.
* Other serious, uncontrolled comorbidities that may affect protocol compliance or interfere with interpretation of results: (1) Active infection or unexplained fever of > 38.5℃ during screening or before first administration (subject fever due to tumor can be included as judged by the investigator); (2) uncontrolled diabetes mellitus; (3) Severe or uncontrolled cardiac clinical symptoms or diseases requiring treatment, such as NYHA Grade II or above heart failure; Unstable angina pectoral; Myocardial infarction occurred within 1 year; Patients with clinically significant supraventricular or ventricular arrhythmias requiring clinical intervention. (4) Pulmonary disease (interstitial pneumonia, obstructive pulmonary disease, and a history of symptomatic bronchospasm).
* Active tuberculosis, hepatitis B (HBV), hepatitis C (HCV) or human immunodeficiency virus (HIV).
* Except for active autoimmune diseases requiring systemic treatment: patients with a history of hypothyroidism who do not need hormone therapy or who are receiving physiological dose hormone replacement therapy; Subjects with stable type 1 diabetes with blood sugar under control.
* Known to be allergic to pemetrexed, nab-paclitaxel, cisplatin, carboplatin or any of their prophylactic agents, or to any of the ingredients of toripalimab.
* An antitumor monoclonal antibody (mAb) received within 4 weeks prior to initial study drug use, or an adverse event from a previous drug that has not recovered (i.e., grade 1 ≤ or at baseline). Note: Except for subjects with grade ≤2 neuropathy or grade ≤2 alopecia, if the subject has undergone major surgery, the toxicity and/or complications resulting from the surgical intervention must be fully recovered before treatment is initiated.
* The live vaccine received within 4 weeks prior to the first use of the study drug is allowed to receive the inactivated virus vaccine for seasonal influenza by injection, but the live attenuated influenza vaccine administered through the nose is not allowed to receive.
* As judged by the Investigator, the subjects have other factors that may cause them to be forced to terminate the study, such as other serious diseases (including mental illness) requiring combined treatment, serious abnormal laboratory test values, family or social factors that may affect the subjects' safety or the data collection of the study.
* Pregnant or lactating women, fertile men and women who were unwilling to use effective contraceptive methods during the study period.
* Other conditions judged by the investigator to be unsuitable for inclusion in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-08-31 (Actual); Primary Completion 2023-08-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Progress Free Survival(PFS) | the time from the date of the operation until the first recurrence or the last follow-up(Up to approximately 26 months).
  Progress Free Survival is defined as included the development of new metastases, or local progression of metastases or primary lesions that underwent surgical resection/radiotherapy and will be assessed according to RESIST 1.1 criteria.

SECONDARY OUTCOMES:
Pathological complete response(pCR) | after 3-4 cycles of neoadjuvant therapy (At the day of surgery)
  Pathological complete response is defined as 0% survival of tumor cells in surgically resected primary and metastatic tumor samples (excluding brain and bone metastases) after neoadjuvant therapy, as assessed by tumor regression grade.
Main pathology rate(MPR) | after 3-4 cycles of neoadjuvant therapy (At the day of surgery)
  Main pathology rate is defined as survival of tumor cells ≤ 10% in surgically resected primary and metastatic tumor samples (excluding brain and bone metastases) after neoadjuvant therapy, assessed by tumor regression grade.
Objective Response Rate (ORR) | after 3-4 cycles of neoadjuvant therapy(Up to approximately 26 months).
  Objective Response Rate is defined as complete response (CR) + partial response (PR), from the beginning of regimental therapy to the end of neoadjuvant therapy, the efficacy of baseline target lesions (primary + metastatic) was assessed by RECIST1.1 criteria.
Assess adverse events | the time from the neoadjuvant until the last follow-up(Up to approximately 26 months).
  Assess all adverse events according to the NCI Common Terminology Criteria for (NCI-CTCAE) v 4.0.3.

CONTACTS AND LOCATIONS:
Overall Officials: Tao Jiang, PH.D, Principal Investigator — The Fourth Military Medical University Tangdu Hospital
Locations (1):
- The Fourth Military Medical University Tangdu Hospital, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No